CLINICAL TRIAL: NCT02103296
Title: Umbilical Cord Blood Use For Admission Blood Tests of Very Low Birth Weight (VLBW) Preterm Neonates: A Multi-center Randomized Clinical Trial
Brief Title: Umbilical Cord Blood Use For Admission Blood Tests of Very Low Birth Weight Preterm Neonates: A Multi-center Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capt Alicia Prescott (U.S. Federal Agency)
Collaborators: C.R.Darnall Army Medical Center (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Capt Alicia Prescott, Associate Investogator, San Antonio Military Medical Center
Organization: San Antonio Military Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 393720-1
Record Dates: First submitted 2014-03-17; First posted 2014-04-03 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant Blood (Active Comparator): Control group. Admission labs to be drawn directly from the infant.
  Interventions: Procedure: Drawing admission labs from infant blood
- Cord Blood (Experimental): Admission labs to be drawn from the infant's cord blood
  Interventions: Procedure: Drawing admission labs from cord blood

INTERVENTIONS:
Procedure: Drawing admission labs from cord blood
  Arms: Cord Blood
Procedure: Drawing admission labs from infant blood
  Arms: Infant Blood

SUMMARY:
The goal of this protocol is to establish a randomized clinical trial comparing the use of cord blood vs. infant blood with the primary outcome of comparing both the absolute hemoglobin concentration and the percent change in hemoglobin concentration from baseline around 24 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than 1200g or Gestational Age less than 30 weeks born at participating medical centers

Exclusion Criteria:

* No specific exclusion criteria

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Absolute hemoglobin concentration | 24 hours of life
Percent change in hemoglobin concentration from baseline | 24 hours of life

SECONDARY OUTCOMES:
Number/volume of packed red blood cell (pRBC) transfusions | Participants will be followed from birth until time of hospital discharge, an expected average of 13 weeks
Number of blood donor exposures | Participants will be followed from birth until time of hospital discharge, an expected average of 13 weeks.
Use of Vasopressors | Participants will be followed from birth until time of hospital discharge, an expected average of 13 weeks.
Hemoglobin concentration at one week of life | one week
Hemoglobin concentration at time of hospital discharge | Approximately 10 - 16 weeks
Head Ultrasound | Read at 7 Days of life and at hospital discharge which is approximately 13 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Thornton S Mu, MD, Principal Investigator — San Antonio Military Medical Center
Locations (6):
- United States (6):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Carl R. Darnall Army medical Center, Fort Hood, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Portsmouth Naval Medical Center, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Derived] Mu TS, Prescott AC, Haischer-Rollo GD, Aden JK, Shapiro JB. Umbilical Cord Blood Use for Admission Blood Tests of VLBW Preterm Neonates: A Randomized Control Trial. Am J Perinatol. 2023 Jul;40(10):1119-1125. doi: 10.1055/s-0041-1733781. Epub 2021 Aug 18. PMID 34407547